CLINICAL TRIAL: NCT05429762
Title: Open-label Study Evaluating the Effect of Tusamitamab Ravtansine on the QTc Interval in Participants With Metastatic Solid Tumors
Brief Title: Effect of Tusamitamab Ravtansine on QTc Interval in Participants With Metastatic Solid Tumors
Acronym: TusaRav-QT
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Tusamitamab ravtansine clinical development program is discontinued as CARMEN-LC03 trial did not meet dual primary endpoint of improving progression-free survival. The decision is not related to any safety concern.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TES16382; U1111-1269-6291 (Registry Identifier: ICTRP); 2022-001213-39 (EudraCT Number)
Record Dates: First submitted 2022-06-08; First posted 2022-06-23 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — tusamitamab ravtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tusamitamab ravtansine (Experimental): Participants will receive tusamitamab ravtansine intravenous (IV) infusion until disease progression, unacceptable toxicity, the start of a new anti-cancer therapy, or the participant's or Investigator's decision to stop the treatment, whichever comes first.
  Interventions: Drug: Tusamitamab ravtansine

INTERVENTIONS:
Drug: Tusamitamab ravtansine — Pharmaceutical form: Concentrated solution for intravenous (IV) administration; Route of administration: IV infusion
  Other Names: SAR408701

SUMMARY:
This is a Phase1, single-arm study for treatment. This is a prospective multicenter, multinational, open-label study to assess the effect of tusamitamab ravtansine on the QT interval in participants with metastatic colorectal cancer (CRC), nonsquamous non small cell lung cancer (NSQ NSCLC), or gastric/ gastroesophageal junction (GEJ) adenocarcinoma for which in the judgement of the Investigator, no standard alternative therapy is available.

DETAILED DESCRIPTION:
This is a single arm study in which participants will receive treatment with tusamitamab ravtansine until disease progression, unacceptable toxicity, the start of a new anti-cancer therapy, or the participant's or Investigator's decision to stop the treatment, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of colorectal cancer (CRC) adenocarcinoma, nonsquamous non small cell lung cancer (NSQ NSCLC), or gastric/ gastroesophageal junction (GC/GEJ) adenocarcinoma, metastatic disease at study entry.
* Participants with documented disease progression, for which, in the judgment of the Investigator, no alternative medical therapy is available.
* Expression of carcinoembryonic antigen-related cell adhesion molecule 5 (CEACAM5) will be assessed centrally using the most recent archival tumor tissue (or, if not available, a fresh biopsy sample) and at least 5 fresh-cut slides of formalin-fixed paraffin embedded (FFPE) tumor tissue sectioned. If less material is available, the participant could still be considered eligible after discussion with the Sponsor.

  * Participants with CRC tumors may be assumed to have adequate CEACAM5 expression without testing results (it will be assessed retrospectively),
  * Participants with NSQ NSCLC must have tumors expressing CEACAM5 or high circulating CEA if tumor tissue is not available.
  * Participants with GC/GEJ must have tumors expressing CEACAM5
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, as determined by the Investigator.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to1.
* A female participant is eligible to participate if she is not pregnant or breastfeeding, is not a woman of childbearing potential (WOCBP) and is a WOCBP and agrees to use a contraceptive method that is highly effective and for at least 7 months after the last dose of treatment. administration.
* Male participant who agrees to use effective contraception methods during and for at least 4 months after the last dose of treatment administration.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Untreated brain metastases that may be considered active or leptomeningeal metastasis. A participant with asymptomatic brain metastasis/metastases is eligible.
* Significant concomitant illness
* History within the last 2 years of an invasive malignancy other than that treated in this study, with the exception of resected/ablated basal or squamous-cell carcinoma of the skin or carcinoma in situ of the cervix, or other local tumors considered cured by local treatment.
* Any major surgery within 3 weeks prior to of first study intervention administration.
* Known uncontrolled infection with human immunodeficiency virus (HIV). Participants with a well-controlled HIV infection/disease must be on antiretroviral therapy (ART) to be eligible.
* Active infection with hepatitis A, B, or C.
* Nonresolution of any prior treatment-related toxicity .
* Unresolved corneal disorder or any previous corneal disorder.
* Use of contact lenses is not permitted.
* Prior history of Torsades de Pointes, or congenital long QT syndrome.
* Patient receives (and cannot discontinue) or is scheduled to receive a QT-prolonging drug unless if deemed necessary for the participant as per the investigators' judgment and started at least 4 weeks prior IMP administration at the same dose and the same frequency.
* QTcF interval >480 msec on screening ECG.
* Poor bone marrow, liver, kidney functions, or electrolytes values
* Participant not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or participants potentially at risk of noncompliance to study procedures.

The above information is not intended to contain all considerations relevant to the potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in QT-interval corrected (QTcF) centrally assessed | Baseline, Cycle 1, and Cycle 2 (1 Cycle = 2 weeks)

SECONDARY OUTCOMES:
Electrocardiogram (ECG) parameter: heart rate (HR) | Baseline, Cycle 1, and Cycle 2 (1 Cycle = 2 weeks)
  To assess the effect of tusamitamab ravtansine (i.e., change from baseline) on cardiac parameters such as heart rate (HR).
ECG parameter: QT interval | Baseline, Cycle 1, and Cycle 2 (1 Cycle = 2 weeks)
  To assess the effect of tusamitamab ravtansine (i.e., change from baseline) on cardiac parameters such as QT interval.
ECG parameter: QT interval corrected according to the Bazett's formula (QTcB) | Baseline, Cycle 1, and Cycle 2 (1 Cycle = 2 weeks)
  To assess the effect of tusamitamab ravtansine (i.e., change from baseline) on cardiac parameters such as QT interval corrected according to the Bazett's formula (QTcB).
ECG parameter: QRS interval | Baseline, Cycle 1, and Cycle 2 (1 Cycle = 2 weeks)
  To assess the effect of tusamitamab ravtansine (i.e., change from baseline) on cardiac parameters such as QRS interval.
ECG parameter: PR interval | Baseline, Cycle 1, and Cycle 2 (1 Cycle = 2 weeks)
  To assess the effect of tusamitamab ravtansine (i.e., change from baseline) on cardiac parameters such as PR interval.
Maximum concentration observed (Cmax) | Multiple timepoint at Cycle 1 (1 Cycle = 2 weeks)
Area under the plasma concentration versus time curve from time 0 to 14 days (AUC0-14d) | Multiple timepoint at Cycle 1 (1 Cycle = 2 weeks)
Incidence of participants with treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and laboratory abnormalities | From the date of first infusion up to approximately 30 days after the last infusion i.e., up approximately 34 weeks
  Assessed according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Overall response rate (ORR) | Up to approximately 30 weeks
  The ORR, defined as the proportion of participants who have a confirmed complete response (CR) or partial response (PR) as the best overall response as determined by investigator/local radiologist review per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) criteria
Duration of response (DOR) | Up to approximately 30 weeks
  The DOR, defined as the time from the first documented evidence of confirmed complete response (CR) or partial response (PR) until progressive disease (PD) as determined by investigator/local radiologist review per RECIST v1.1 criteria or death (due to any cause), whichever comes first

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (7):
- Mary Crowley Cancer Research Center Site Number : 8400002, Dallas, Texas, United States
- Investigational Site Number : 0560001, Edegem, Belgium
- France (2):
  - Investigational Site Number : 2500001, Dijon
  - Investigational Site Number : 2500002, Marseille
- Spain (2):
  - Investigational Site Number : 7240002, Barcelona, Catalunya [Cataluña]
  - Investigational Site Number : 7240001, Madrid, Madrid, Comunidad de
- Investigational Site Number : 7920001, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: TES16382 Plain language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25363&tenant=MT_SNY_9011